CLINICAL TRIAL: NCT01315236
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Liposomal Amikacin for Inhalation in Patients With Recalcitrant Nontuberculous Mycobacterial Lung Disease
Brief Title: Liposomal Amikacin for Inhalation (LAI) for Nontuberculous Mycobacteria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR02-112
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Mycobacterium Infections, Nontuberculous
Keywords: Amikacin Liposome Inhalation Suspension (ALIS); Arikayce
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAI 590 mg QD (Experimental): LAI 590 mg QD
  Interventions: Drug: Liposomal amikacin for inhalation (LAI)
- Placebo (Placebo Comparator): placebo QD
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Liposomal amikacin for inhalation (LAI) — * Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * Liposomal amikacin for inhalation will be administered for 84 days in the double-blind, randomized portion of the study.
  * Subjects can continue with 84 additional days of dosing in the open label extension.
  Other Names: Amikacin Liposome Inhalation Suspension (ALIS); Arikayce
  Arms: LAI 590 mg QD
Drug: placebo — * Placebo is provided as a sterile aqueous lipid dispersion for inhalation via nebulization.
  * Administration procedures, volume and administration time are similar to LAI.
  * Placebo will be administered for 84 days only during the double-blind, randomized portion of the study.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of 84 days of daily dosing of 590 mg of LAI versus placebo in patients with treatment refractory NTM lung disease.

The first part of the study is the 84-day double-blind phase to evaluate the primary and secondary endpoints.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, double-blind study of efficacy, safety, and tolerability of once daily (QD) dosing of LAI 590 mg versus placebo for 84 days in subjects with treatment refractory NTM lung infection on a stable multidrug regimen. At the conclusion of the randomized double-blind phase of the study, subjects who consented to continue in the open-label phase of the study received LAI 590 mg QD for 84 additional days. All subjects were required to complete a 28-day safety follow-up after their end of treatment study visit (Day 168). Subjects completing this study were consented for enrollment in a long-term follow-up phase and were asked to return to the study site at 12 months and 24 months (per protocol Amendment #3, the 24-month follow-up visit was no longer required) (visit window ± 2 months) after the last dose of study drug (either after completing the randomized double-blind phase or the open-label phase). Subjects were stratified upon entering the study based on the presence or absence of cystic fibrosis (CF) and Mycobacterium avium complex versus M abscessus as the predominate NTM organism at baseline and were block randomized to receive either LAI or placebo in a 1:1 ratio in the double-blind phase.

Subjects completing the main study, and subjects who completed the 84-day open-label phase, were consented for enrollment in a post-LAI safety follow-up assessment and were asked to return to the study site 12 months (visit window ± 2 months) after the last dose of study drug (either after completing the randomized double-blind phase or the open-label phase). The screening period required obtaining 3 morning sputum specimens (spontaneous or induced) for mycobacteriology. At each post-screening sputum timepoint, at least 2 and preferably 3 sputum specimens were obtained. At Day 1 (baseline), subjects were evaluated pre-dose and post-dose at the study site. Subjects returned to the study site briefly on Day 2 for collection of serum samples to determine creatinine clearance. On Days 28, 56, and 84, study drug was administered at the site and the efficacy, safety, and tolerability of study drug were evaluated. At Day 85, those subjects continuing in the open-label phase of the study received LAI 590 mg at the study site with pre-dose and post-dose assessments for safety and efficacy. Subjects returned every 28 days (Days 112, 140, and 168) in the open-label phase. A 28-day, post-dose follow-up visit occurred at either Day 112 for those subjects who did not continue in the open-label phase or at Day 196 for those subjects who continued in the open-label phase.

Subjects completing the main study, and subjects who completed the 84-day open-label phase, were consented for enrollment in a post-LAI safety follow-up assessment and were asked to return to the study site 12 months (visit window ± 2 months) after the last dose of study drug (either after completing the randomized double-blind phase or the open-label phase). Arikace™, Arikayce™, Liposomal Amikacin for Inhalation (LAI), and Amikacin Liposome Inhalation Suspension (ALIS) may be used interchangeably throughout this study and other studies evaluating amikacin liposome inhalation suspension.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of pulmonary nontuberculous mycobacterial lung disease in accordance with the 2007 ATS/IDSA criteria with evidence of nodular bronchiectasis and/or cavitary disease by chest computed tomography (CT).
2. History of chronic infection with either Mycobacterium avium complex or Mycobacterium abscessus or mixed infection with both species (defined as at least 2 documented positive cultures in the prior 2 years, of which at least one was obtained in the 6 months prior to screening).
3. Positive sputum culture obtained at screening visit with either Mycobacterium avium complex or Mycobacterium abscessus or mixed infection with one dominant species.
4. Receiving ATS/IDSA guidelines-based treatment regimen defined as: adherent to a multi-drug regimen for at least 6 months prior to screening with persistently positive mycobacterial cultures.
5. Ability to produce at least 3 mL of sputum or be willing to undergo an induction that produces at least 3 mL of sputum for clinical evaluation.
6. Female of childbearing potential agrees to practice an acceptable method of birth control (e.g., abstinence, hormonal or barrier methods, partner sterilization, or IUD).

Key Exclusion Criteria:

1. Forced Expiratory Volume in 1 second (FEV1) <30% of predicted at Screening.
2. Presence of any clinically significant cardiac disease as determined by Investigator. The QTc criteria for Exclusion is QTc> 450 msec for males or QTc> 470 msec for females.
3. Subjects with hemoptysis of ≥60 mL in a 24 hour period within 4 weeks prior to screening.
4. Active pulmonary malignancy (primary or metastatic) or any malignancy requiring chemotherapy or radiation therapy within one year prior to screening or anticipated during the study period.
5. Active allergic bronchopulmonary mycosis or any other condition requiring systemic steroids at a dose > equivalent of 10 mg/day of prednisone within 3 months prior to screening or anticipated during the study period.
6. Pulmonary tuberculosis requiring treatment or treated within 2 years prior to screening.
7. History of lung transplantation.
8. Hypersensitivity to aminoglycosides.
9. Any change in chronic NTM multi-drug regimen within 28 days prior to Study Day 1.
10. Evidence of biliary cirrhosis with portal hypertension.
11. History of daily, continuous oxygen supplementation.
12. Smoking tobacco or any substance within 6 months prior to screening or anticipated inability to refrain from smoking throughout the study.

Subjects with CF or primary ciliary dyskinesia were eligible to participate in the study if all eligibility criteria defined above were met. Subjects with CF were required to have documented confirmation of CF to be eligible for the study. The CF diagnosis had to be documented by a positive sweat test ≥ 60 mmol/L or by DNA analysis revealing both mutated alleles consistent with CF disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-04-19 (Actual); Primary Completion 2014-08-18 (Actual); Study Completion 2015-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Eagle, Study Director — Insmed Incorporated
Locations (19):
- United States (18):
  - Birmingham, Alabama
  - Stanford, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Tampa, Florida
  - Kansas City, Kansas
  - Bethesda, Maryland
  - Rochester, Minnesota
  - New York, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Tyler, Texas
  - Milwaukee, Wisconsin
- Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Rubino CM, Onufrak NJ, van Ingen J, Griffith DE, Bhavnani SM, Yuen DW, Mange KC, Winthrop KL. Population Pharmacokinetic Evaluation of Amikacin Liposome Inhalation Suspension in Patients with Treatment-Refractory Nontuberculous Mycobacterial Lung Disease. Eur J Drug Metab Pharmacokinet. 2021 Mar;46(2):277-287. doi: 10.1007/s13318-020-00669-7. Epub 2021 Feb 17. PMID 33595792
- [Derived] Olivier KN, Griffith DE, Eagle G, McGinnis JP 2nd, Micioni L, Liu K, Daley CL, Winthrop KL, Ruoss S, Addrizzo-Harris DJ, Flume PA, Dorgan D, Salathe M, Brown-Elliott BA, Gupta R, Wallace RJ Jr. Randomized Trial of Liposomal Amikacin for Inhalation in Nontuberculous Mycobacterial Lung Disease. Am J Respir Crit Care Med. 2017 Mar 15;195(6):814-823. doi: 10.1164/rccm.201604-0700OC. PMID 27748623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One patient out of the 90 was randomized but not dosed.
Groups:
- LAI 590 mg QD: LAI 590 mg QD
  Liposomal amikacin for inhalation (LAI): - Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * Liposomal amikacin for inhalation will be administered for 84 days in the double-blind, randomized portion of the study.
  * Subjects can continue with 84 additional days of dosing in the open label extension.
- Placebo: placebo QD
  placebo: - Placebo is provided as a sterile aqueous lipid dispersion for inhalation via nebulization.
  * Administration procedures, volume and administration time are similar to LAI.
  * Placebo will be administered for 84 days only during the double-blind, randomized portion of the study.
Period: Double-blind Phase
Arm/Group | LAI 590 mg QD | Placebo
Started | 44 | 45
Completed | 40 | 45
Not Completed | 4 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal of Consent | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Open-label Phase
Arm/Group | LAI 590 mg QD | Placebo
Started | 35 (Some subjects did not consent to the open label after the double blind phase.) | 43 (Some subjects did not consent to the open label after the double blind phase.)
Completed | 34 | 41
Not Completed | 1 | 2
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Other | 0 | 1
Period: 12-Month Follow-up Period
Arm/Group | LAI 590 mg QD | Placebo
Started | 27 (Some subjects did not consent to the 12 month safety.) | 32 (Some subjects did not consent to the 12 month safety.)
Completed | 26 | 31
Not Completed | 1 | 1
Not completed — Death | 0 | 1
Not completed — Did not return to the site for Month 12 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Double-blind Phase
Groups:
- Total: Total of all reporting groups
Arm/Group | LAI 590 mg QD | Placebo | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (16.61) | 59.1 (15.20) | 58.5 (15.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (not of Hispanic origin) | 42 | 40 | 82
  Hispanic | 0 | 2 | 2
  African | 0 | 1 | 1
  Asian | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Semi-Quantitative Mycobacterial Culture Results From Baseline to Day 84.
Description: The endpoint used the 7-step semi-quantitative scale (SQS) for mycobacterial culture reporting in both solid and liquid growth media, with step 1 = culture negative in both solid and liquid media, step 2 = growth in liquid medium only, 3 = solid medium positive, 4 = 50 to 100 colonies in solid medium & growth in liquid, 5 = >100 to 200 colonies in solid medium & growth in liquid, 6 = >200 to 500 colonies in solid medium & growth in liquid, 7 = >500 colonies in solid medium & growth in liquid. Full scale range is 1 (best score) to 7 (worst score). The change in step measures the growth at Day 84 compared to the growth at Baseline. The negative values represent reduction in colony growth.
Time Frame: Baseline and end of double-blind phase of 84 days
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD | Placebo
Number analyzed (Participants) | 44 | 45
Participants
  Baseline: Culture negative | 5 | 5
  Baseline: Growth in liquid medium only | 1 | 1
  Baseline: Agar positive | 17 | 10
  Baseline: 1+ (50-100 colonies) | 2 | 4
  Baseline: 2+ (> 100-200 colonies) | 2 | 2
  Baseline: 3+ (> 200-500 colonies) | 3 | 4
  Baseline: 4+ (> 500 colonies) | 14 | 19
  Day 84: -6 steps from baseline | 1 | 0
  Day 84: -5 steps from baseline | 0 | 0
  Day 84: -4 steps from baseline | 1 | 0
  Day 84: -3 steps from baseline | 3 | 0
  Day 84: -2 steps from baseline | 6 | 6
  Day 84: -1 step from baseline | 5 | 5
  Day 84: no change from baseline | 23 | 23
  Day 84: +1 step from baseline | 2 | 5
  Day 84: +2 steps from baseline | 0 | 3
  Day 84: +3 steps from baseline | 1 | 0
  Day 84: +4 steps from baseline | 1 | 2
  Day 84: +5 steps from baseline | 0 | 1
  Day 84: +6 steps from baseline | 0 | 0
  Day 84: +7 (Death) | 1 | 0
Statistical Analysis 1: Comparison: LAI 590 mg QD vs Placebo; The primary efficacy analysis tested the following hypotheses: * H0: There is no difference at Day 84 between the LAI arm and the placebo arm * Ha: There is a difference at Day 84 between the LAI arm and the placebo arm Statistical analysis applies to all day 84 rows; Test type: Superiority; p = 0.072, Wilcoxon rank sum test — Conducted in the mITT population using a stratified Wilcoxon rank sum test, to compare the treatment arms at a 2-sided significance level of 0.05, adjusting for the randomization strata (presence/absence of CF and MAC versus Mycobacterium abscessus)

2. Secondary Outcome: Number of Subjects With Negative NTM Culture for the LAI Arm at Day 84 Compared to the Placebo Arm at Day 84
Description: Sputum specimens were cultured in liquid media in addition to solid media (agar). If results were negative on agar, the liquid media was held for 6 weeks before reporting as culture negative. Culture was negative when confirmed with no growth in liquid medium.
Time Frame: 84 days double-blind phase
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD | Placebo
Number analyzed (Participants) | 44 | 45
Participants | 14 | 4
Statistical Analysis 1: Comparison: LAI 590 mg QD vs Placebo; stratified Cochran-Mantel-Haenszel test; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel

3. Secondary Outcome: Time to Negative NTM Culture….During the 84-day Double-blind Treatment Phase
Description: as for outcome 2
Time Frame: 84 days double-blind phase
Population: mITT
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | LAI 590 mg QD | Placebo
Number analyzed (Participants) | 44 | 45
days | NA [85.0 to NA] — The median time to a negative NTM culture was not able to be estimated due to insufficient number of participants. | NA [NA to NA] — The median time to a negative NTM culture was not able to be estimated due to insufficient number of participants.
Statistical Analysis 1: Comparison: LAI 590 mg QD vs Placebo; Cox proportional hazard model; Test type: Superiority; p = 0.0129, Regression, Cox; Cox Proportional Hazard = 5.68, 95% CI 2-sided [1.25 to 25.79]

4. Secondary Outcome: Ordinal, 3-level Response From Baseline on the SQS for Mycobacterial Culture for the LAI Arm at Day 84 Compared to the Placebo Arm at Day 84
Description: The ordinal, 3-level response are (1) improvement (2) no change (3) worsening or death
Time Frame: Baseline and end of double-blind phase of 84 days
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD | Placebo
Number analyzed (Participants) | 44 | 45
Participants
  Improvement (a decrease of 1 step or more) | 16 | 11
  No change | 20 | 23
  Worsening (an increase of 1 step or more) or death | 5 | 11
Statistical Analysis 1: Comparison: LAI 590 mg QD vs Placebo; Ordinal Logistic Regressions Model; Test type: Superiority; p = 0.077, Regression, Logistic

5. Secondary Outcome: Change From Baseline in Respiratory and Systemic Symptoms Questionnaire (RSSQ) Score at Day 84 for the LAI Arm Compared to the Placebo Arm
Description: The RSSQ was administered to gather information from the subject about the types of symptoms that the subject has experienced since the last contact. A reduction in score indicates improvement. The range of values for the scores are -2 (best) to +2 (worst) in whole numbers. The composite score was calculated by averaging the scores of the subscales.
Time Frame: Baseline to day 84.
Population: mITT
Measure: Mean (Standard Deviation); unit: units on a score
Arm/Group | LAI 590 mg QD | Placebo
Number analyzed (Participants) | 44 | 45
units on a score | -0.80 (0.992) | -0.60 (0.736)
Statistical Analysis 1: Comparison: LAI 590 mg QD vs Placebo; Stratified Wilcoxon-rank sum; Test type: Superiority; p = 0.4545, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change From Baseline in Global Rating of Health (GRH) at Day 84 for the LAI Arm Compared to the Placebo Arm
Description: The assessing physician asked the subject to rate his/her assessment of health according to the GRH. Subject responses to, "How would you rate your health at the present time?" included: Excellent, Good, Fair, or Poor.
Time Frame: Baseline and end of double-blind phase of 84 days
Population: mITT
  Subjects with missing data were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | LAI 590 mg QD | Placebo
Number analyzed (Participants) | 44 | 45
Participants
  No change: Excellent -> Excellent: number analyzed (Participants) | 39 | 45
  No change: Excellent -> Excellent | 2 | 2
  No change: Good -> Good: number analyzed (Participants) | 39 | 45
  No change: Good -> Good | 15 | 21
  No change: Fair -> Fair: number analyzed (Participants) | 39 | 45
  No change: Fair -> Fair | 8 | 5
  No change: Poor -> Poor: number analyzed (Participants) | 39 | 45
  No change: Poor -> Poor | 1 | 1
  Increase: number analyzed (Participants) | 39 | 45
  Increase | 4 | 6
  Increase: By 3 Categories (Poor -> Excellent): number analyzed (Participants) | 39 | 45
  Increase: By 3 Categories (Poor -> Excellent) | 0 | 0
  Increase by 2 Categories: number analyzed (Participants) | 39 | 45
  Increase by 2 Categories | 0 | 1
  Increase: By 2 Categories (Poor -> Good): number analyzed (Participants) | 39 | 45
  Increase: By 2 Categories (Poor -> Good) | 0 | 0
  Increase: By 2 Categories (Fair -> Excellent): number analyzed (Participants) | 39 | 45
  Increase: By 2 Categories (Fair -> Excellent) | 0 | 1
  Increase by 1 Category: number analyzed (Participants) | 39 | 45
  Increase by 1 Category | 4 | 5
  Increase: By 1 Category (Poor -> Fair): number analyzed (Participants) | 39 | 45
  Increase: By 1 Category (Poor -> Fair) | 2 | 0
  Increase: By 1 Category (Fair -> Good): number analyzed (Participants) | 39 | 45
  Increase: By 1 Category (Fair -> Good) | 2 | 5
  Increase: By 1 Category (Good -> Excellent): number analyzed (Participants) | 39 | 45
  Increase: By 1 Category (Good -> Excellent) | 0 | 0
  Decrease: number analyzed (Participants) | 39 | 45
  Decrease | 9 | 10
  Decrease: By 3 Categories (Excellent --> Poor): number analyzed (Participants) | 39 | 45
  Decrease: By 3 Categories (Excellent --> Poor) | 0 | 0
  Decrease: By 2 Categories: number analyzed (Participants) | 39 | 45
  Decrease: By 2 Categories | 0 | 0
  Decrease: By 2 Categories (Excellent -> Fair): number analyzed (Participants) | 39 | 45
  Decrease: By 2 Categories (Excellent -> Fair) | 0 | 0
  Decrease: By 2 Categories (Good -> Poor): number analyzed (Participants) | 39 | 45
  Decrease: By 2 Categories (Good -> Poor) | 0 | 0
  Decrease: By 1 Category: number analyzed (Participants) | 39 | 45
  Decrease: By 1 Category | 9 | 10
  Decrease: By 1 Category (Excellent -> Good): number analyzed (Participants) | 39 | 45
  Decrease: By 1 Category (Excellent -> Good) | 2 | 0
  Decrease: By 1 Category (Good -> Fair): number analyzed (Participants) | 39 | 45
  Decrease: By 1 Category (Good -> Fair) | 5 | 7
  Decrease: By 1 Category (Fair -> Poor): number analyzed (Participants) | 39 | 45
  Decrease: By 1 Category (Fair -> Poor) | 2 | 3

7. Secondary Outcome: Number of Participants Requiring "Rescue" Anti-mycobacterial or Other "Rescue" Drugs During the 84-day Double-blind Phase
Description: Per the study protocol, study subjects were on a stable, multi-drug, anti-mycobacterial regimen based on the 2007 ATS/IDSA Guidelines; the regimen should not have changed during the study period except for safety concerns. The need for changes to the concurrent anti-mycobacterial regimen or "rescue" therapy was at the discretion of the Investigator and was tracked as a study outcome.
Time Frame: 84 days double-blind phase
Population: mITT
Measure: Number; unit: participants
Arm/Group | LAI 590 mg QD | Placebo
Number analyzed (Participants) | 44 | 45
participants | 21 | 11
Statistical Analysis 1: Comparison: LAI 590 mg QD vs Placebo; Cox Proportional Hazard Model; Test type: Superiority; p = 0.0076, Regression, Cox; Cox Proportional Hazard = 2.69, 95% CI 2-sided [1.28 to 5.64]

8. Secondary Outcome: Number of Subject for "Rescue" Anti-mycobacterial or Other "Rescue" Drugs During the 84-day Double-blind Phase
Description: as for outcome 7
Time Frame: 84 days double-blind phase
Population: mITT
Measure: Number; unit: participants
Arm/Group | LAI 590 mg QD | Placebo
Number analyzed (Participants) | 44 | 45
participants
  Number of subjects with the event | 21 | 11
  Number censored | 23 | 34

ADVERSE EVENTS:
Time Frame: Up to Day 196 (84 days double-blind phase + 84 days open label phase + 28 days post discontinuation of study drug). Adverse events (AEs) were not collected during the 12-month follow-up period..
Groups:
- LAI 590 mg QD - Double Blind: LAI 590 mg QD
  Liposomal amikacin for inhalation (LAI): - Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * Liposomal amikacin for inhalation will be administered for 84 days in the double-blind, randomized portion of the study.
  * Subjects can continue with 84 additional days of dosing in the open label extension.
- Placebo - Double Blind: placebo QD
  placebo: - Placebo is provided as a sterile aqueous lipid dispersion for inhalation via nebulization.
  * Administration procedures, volume and administration time are similar to LAI.
  * Placebo will be administered for 84 days only during the double-blind, randomized portion of the study.
- LAI 590 mg QD - Open Label: LAI 590 mg QD
  Liposomal amikacin for inhalation (LAI): - Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  - 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  Subjects can continue with 84 additional days of dosing in the open label extension.
- Placebo - Open Label: placebo QD
  placebo: - Placebo is provided as a sterile aqueous lipid dispersion for inhalation via nebulization.
  Subjects can continue with 84 additional days of dosing in the open label extension.
Arm/Group | LAI 590 mg QD - Double Blind | Placebo - Double Blind | LAI 590 mg QD - Open Label | Placebo - Open Label
All-Cause Mortality (participants affected / at risk) | 1/44 | 0/45 | 1/35 | 0/43
Serious Adverse Events (participants affected / at risk) | 8/44 | 4/45 | 5/35 | 5/43
Other Adverse Events (participants affected / at risk) | 41/44 | 39/45 | 31/35 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAI 590 mg QD - Double Blind (N=44) | Placebo - Double Blind (N=45) | LAI 590 mg QD - Open Label (N=35) | Placebo - Open Label (N=43)
Infective exacerbation of bronchiectasis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAI 590 mg QD - Double Blind (N=44) | Placebo - Double Blind (N=45) | LAI 590 mg QD - Open Label (N=35) | Placebo - Open Label (N=43)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 3 (3) | 5 (6)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (5)
Fatigue (General disorders) | 7 (8) | 4 (4) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 3 (6) | 3 (4) | 1 (1)
Chest discomfort (General disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 17 (21) | 9 (9) | 9 (9) | 15 (16)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 (3) | 1 (1) | 4 (5) | 6 (8)
Laryngitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (7) | 2 (2) | 5 (5)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 19 (25) | 4 (4) | 3 (3) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 6 (6) | 3 (3) | 8 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1) | 3 (6) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6) | 5 (5) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (2) | 0 (0) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the signed Investigator Agreement in the protocol and protocol amendments, the PI agreed that the information presented in the study protocol is confidential, and assured that no information based on the conduct of the study was released without prior Insmed Incorporated Consent, unless the requirement is superseded by the Food and Drug Administration or other regulatory authority.